CLINICAL TRIAL: NCT07193004
Title: Quality of Life Improvement After Transcatheter Aortic Valve Implantation (TAVI) in the UK: A Prospective 1-Year Study (QualiTAVI-UK Trial)
Brief Title: Quality of Life Improvement After TAVI (QualiTAVI-UK Trial)
Acronym: QualiTAVI-UK
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Principal Investigator, Ayman Helal, Professor, University Hospital Plymouth NHS Trust
Other Study IDs: 25/CAR/222
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: TAVI(Transcatheter Aortic Valve Implantation); TAVI; Quality of Life; Mental Health
Keywords: Transcatheter aortic valve implantation (TAVI); quality of life; Kansas City Cardiomyopathy Questionnaire; Mini-Montreal Cognitive Assessment (Mini-MoCA); life expectancy; Mental health; Clinical Frailty Scale (CFS)
MeSH Terms: conditions — Psychological Well-Being | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAVI: Patients who were eligible and accepted for TAVI procedure regardless of the patient's age and informed consent provided by the patient for the TAVI procedure.
  Interventions: Behavioral: Quality of Life

INTERVENTIONS:
Behavioral: Quality of Life — Measures - We will use the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) to assess QoL, Mini-Montreal Cognitive Assessment (Mini-MoCA) to assess cognitive function, the Clinical Frailty Scale (CFS) to assess frailty status, and life expectancy estimation by the heart team to categorize patients as having: 1-2 years expected survival or more than 2 years expected survival (This will allow for an analysis of how life expectancy correlates with QoL improvements after TAVI).
  Assessment Timeline - Patients will be assessed at four key time points: at time of referral (baseline assessment), pre-procedure (to assess impact of delay on the patient), 30 days post-TAVI (early follow-up to assess recovery and improvement in QoL), and 3 months post-TAVI (longer-term follow-up to evaluate sustained QoL changes). At each time point, the KCCQ-12, Mini-MoCA, and Clinical Frailty Scale (CFS) will be administered.
  Other Names: KCCQ-12; CFS; Mini-MoCA

SUMMARY:
Transcatheter aortic valve implantation (TAVI) has become an important therapeutic intervention for patients with symptomatic severe aortic stenosis (AS) who are at high surgical risk. While the clinical outcomes of TAVI are well established, there is limited data on the long-term quality of life (QoL) following the procedure. This prospective study will assess QoL in patients undergoing TAVI at Derriford Hospital, University Hospitals Plymouth, UK. Investigators will employ the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) and Mini-Montreal Cognitive Assessment (Mini-MoCA) to evaluate both physical and mental health outcomes, supplemented by an analysis of life expectancy estimated by a multidisciplinary team (MDT). Data will be collected at referral, pre-procedural, 30 days, and 3 months post-TAVI. This will be the first prospective trial focused on QoL improvement after TAVI, as all previous studies have been retrospective in nature. The study aims to provide comprehensive insights into the QoL improvements after TAVI, which will guide future clinical decision-making in this population.

DETAILED DESCRIPTION:
Study Title uality of Life Improvement after Transcatheter Aortic Valve Implantation (TAVI) in the UK: A Prospective 1-Year Study (QualiTAVI-UK trial)

Study Design This is a prospective, single-center study that will be conducted over 1 year at Derriford Hospital, University Hospitals Plymouth, UK.

Study Participants The study will include all patients undergoing TAVI for severe AS during this period.

Eligibility Criteria Inclusion Criteria: Patients who were eligible and accepted for TAVI procedure regardless of the patient's age and informed consent provided by the patient for the TAVI procedure.

Exclusion Criteria: Patients who declined enrollment in this research.

Planned Sample Size More than 100 patients

Follow-up Duration 3 months

Planned Study Period 1 year

Primary Objective This study aims to address the knowledge gap regarding the impact of TAVI on Quality of Life (QoL) Secondary Objective -

ELIGIBILITY:
Inclusion Criteria:

* Patients who were eligible and accepted for TAVI procedure regardless of the patient's age and informed consent provided by the patient for the TAVI procedure.

Exclusion Criteria:

* Patients who declined enrollment in this research.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were eligible and accepted for TAVI procedure regardless of the patient's age and informed consent provided by the patient for the TAVI procedure.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of QoL | 30 days post-TAVI (early follow-up to assess recovery and improvement in QoL), and 3 months post-TAVI
  This is defined as improvement in QoL scores from baseline to 3 months post-TAVI. Based on KCCQ-12, a change of 5 points (small but clinically important change), 10 points (moderate-to-large), and 20 points (large-to-very large clinical changes). Based on CFS score, worsened frailty is defined as an increase in CFS score of +4, and improved frailty by a decrease of -2.

SECONDARY OUTCOMES:
Correlation between life expectancy and QoL improvements | 30 days post-TAVI (early follow-up to assess recovery and improvement in QoL), and 3 months post-TAVI
  Correlation between life expectancy and QoL improvements using regression analysis. Mental health and cognitive function (Mini-MoCA scores), frailty status (CFS), will be explored as potential mediators of QoL outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Helal, MD Cardiology, Study Chair — University Hospitals Plymouth NHS Trust; Ayman Helal, MD Cardiology, Principal Investigator — University Hospitals Plymouth NHS Trust
Locations (1):
- Derriford Hospital, Plymouth, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Relevant information related to the study will be shared

REFERENCES:
- [Background] Monnin C, Besutti M, Ecarnot F, Guillon B, Chatot M, Chopard R, Yahia M, Meneveau N, Schiele F. Prevalence and severity of cognitive dysfunction in patients referred for transcatheter aortic valve implantation (TAVI): clinical and cognitive impact at 1 year. Aging Clin Exp Res. 2022 Aug;34(8):1873-1883. doi: 10.1007/s40520-022-02102-2. Epub 2022 Mar 11. PMID 35275374
- [Background] Shimura T, Yamamoto M, Kano S, Kagase A, Kodama A, Koyama Y, Tsuchikane E, Suzuki T, Otsuka T, Kohsaka S, Tada N, Yamanaka F, Naganuma T, Araki M, Shirai S, Watanabe Y, Hayashida K; OCEAN-TAVI Investigators. Impact of the Clinical Frailty Scale on Outcomes After Transcatheter Aortic Valve Replacement. Circulation. 2017 May 23;135(21):2013-2024. doi: 10.1161/CIRCULATIONAHA.116.025630. Epub 2017 Mar 16. PMID 28302751
- [Background] Kennon S, Styra R, Bonaros N, Stastny L, Romano M, Lefevre T, Di Mario C, Stefano P, Ribichini FL, Himbert D, Urena-Alcazar M, Salgado-Fernandez J, Cuenca Castillo JJ, Garcia B, Deutsch C, Sykorova L, Kurucova J, Thoenes M, Luske C, Bramlage P, Frank D. Quality of life after transcatheter or surgical aortic valve replacement using the Toronto Aortic Stenosis Quality of Life Questionnaire. Open Heart. 2021 Nov;8(2):e001821. doi: 10.1136/openhrt-2021-001821. PMID 34810276